CLINICAL TRIAL: NCT03748524
Title: Washington University (WU) 321: Analysis of Antigen Specific B Cell Responses to Immunization With Influenza Virus Vaccine: Fine Needle Aspiration (FNA) and Bone Marrow Aspiration (BMA)
Brief Title: Analysis of Antigen Specific B Cell Responses to Immunization With Influenza Virus Vaccine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201808171
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Immunity, Cellular
Keywords: Influenza, B cells, Antibodies, Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Influenza Vaccine (Experimental): Single Influenza Vaccine,Quadrivalent
  Interventions: Drug: Influenza Vaccine

INTERVENTIONS:
Drug: Influenza Vaccine — Influenza Vaccine,Quadrivalent SIngle vaccination all participants at day 0

SUMMARY:
Immunization with the inactivated influenza vaccine with blood samples collected at 7 visits (baseline, day 7, 14, 28, 60, 90 and 180, fine needle aspiration (FNAs) from axillary lymph nodes at baseline, days, 4, 14, 28, 60 and 180. BMA at baseline, days 28 and 180.

DETAILED DESCRIPTION:
IM Immunization with the inactivated influenza vaccine with blood samples collected at 7 visits (baseline, day 7, 14, 28, 60, 90 and 180, fine needle aspiration (FNAs) from axillary lymph nodes at baseline, days, 4, 14, 28, 60 and 180. BMA at baseline, days 28 and 180.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give informed consent
2. Capable of attending all study visits according to the study schedule.
3. Males or females between the ages of 18 to 50 (inclusive).
4. Are in good health, as determined by medical history and targeted physical exam related to this history.
5. Participants agree not to take any vaccines in the first 60 days after receipt of the influenza vaccine
6. The following laboratory values obtained within 14 days prior to entry..

   * Absolute neutrophil count (ANC) ≥750 cells/mm3
   * Hemoglobin ≥11.0 g/dL for men and ≥10.0 g/dL for women
   * Platelet count ≥100,000/mm3
   * Creatinine clearance ≥60 mL/min estimated by the Cockcroft-Gault equation
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (SGPT) ≤5.0 times upper limit of normal (ULN)
7. Willing to:

   * give FNA specimens for the study. (even if he/she are not willing to give bone marrow aspirates (for any reason), they can be enrolled)
   * give bone marrow aspirates, but we cannot locate axillary lymph nodes
   * give both FNA and BMA specimens

Exclusion Criteria:

* 1. History influenza vaccination for the last three years.

  2. Coagulopathy (primary or iatrogenic) which would contraindicate FNA

  3. Any history of allergy to eggs, chicken or gelatin or to any previous influenza vaccine

  4. Have an acute illness within 72 hours before vaccination.

  5. A history of a medical condition resulting in impaired immunity (such as HIV infection, cancer, particularly leukemia, lymphoma, use of immunosuppressive or antineoplastic drugs or X-ray treatment). Persons with previous skin cancers or cured non-lymphatic tumors are not excluded from the study.

  6. History of HIV infection, Hepatitis B or Hepatitis C infection

  7. History of any chronic medical conditions that are considered progressive (ex, diabetes, heart disease, lung disease, liver disease, kidney disease, gastrointestinal diseases and uncontrolled hypertension).

  8. History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the study.

  9. Have taken oral or parenteral corticosteroids of any dose within 30 days before study vaccination.

  10. Have taken high-dose inhaled corticosteroids within 30 days before study vaccination.

  11. Autoimmune disorders; mild autoimmune disorders such as eczema is not exclusion after assessment by the investigator.

  12. Recipient of a blood products or immune globulin product within 42 days of the vaccination visit.

  13. Pregnant women and nursing mothers or women who are planning to become pregnant for the study duration.

  14. Have received any licensed live vaccine within 30 days or any licensed inactivated vaccine within 14 days prior to study vaccination.

  15. Have planned vaccination with any vaccine during first 60 days of study participation.

  16. Have received immunoglobulin or other blood products, with the exception of Rho D immunoglobulin, within 90 days prior to study vaccination.

  17. Have donated blood or blood products within 30 days before study vaccination, plan to donate blood at any time during the duration of subject study participation, or plan to donate blood within 30 days after the last blood draw.

  18. Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of subjects achieving seroconversion | 0 and day 28
  Change in serum hemagglutination-inhibition (HAI) antibody titers between day 0 to day 28

SECONDARY OUTCOMES:
Determine the frequency of vaccine-induced responses | Day7
  Frequency of vaccine-specific plasmablasts detected in blood at day 7 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ellebedy, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Infectious Disease Clinical Research Unit, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No